CLINICAL TRIAL: NCT02724618
Title: Phase II Study of Nanocurcumin Versus Placebo for Patients Undergoing Radiotherapy for Prostate Cancer
Brief Title: Nanocurcumin for Prostate Cancer Patients Undergoing Radiotherapy (RT)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Behnam Daheshpour Charity Organization, Tehran, Iran (Unknown)
Responsible Party: Principal Investigator, Bahram Mofid, Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 406
Record Dates: First submitted 2016-03-09; First posted 2016-03-31 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: Curcumin; Protection, Radiation; Controlled Clinical Trials, Randomized; Radiation Therapy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin plus RT (Experimental): 120mg/day nanocurcumin during RT course
  Interventions: Drug: Curcumin; Radiation: RT
- Placebo plus RT (Placebo Comparator): 120mg/day placebo of nanocurcumin during RT course
  Interventions: Radiation: RT; Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — 120mg/d oral nanocurcumin (3 capsules of SinaCurcumin®40 per day) 3 days before and during radiotherapy
  Other Names: SinaCurcumin®
  Arms: Curcumin plus RT
Radiation: RT — EBRT is delivered as Intensity-Modulated Radiation Therapy (IMRT) or 3D-conformal RT
  Other Names: External Beam Radiation Therapy (EBRT)
Drug: Placebo — Placebo (3 placebo capsules of SinaCurcumin®40 per day), 3 days before and during radiotherapy
  Other Names: SinaCurcumin® placebo
  Arms: Placebo plus RT

SUMMARY:
There is a growing body of evidence exploring the role of curcumin as a radioprotector against radiation-induced injury in normal tissues as well as a radiosensitizer in tumor cells. The aim of this study is to determine the efficacy of oral nanocurcumin in prostate cancer patients undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Candidate for External Beam Radiotherapy
* ECOG performance status 0-2

Exclusion Criteria:

* Patients with Metastatic Prostate Cancer
* Patients with Kidney & Liver dysfunction
* Gastrointestinal disorders such as IBD, reflux and peptic ulcers
* Any adverse reaction to curcumin

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Proctitis [assessed using Common terminology criteria for adverse events (CTCAE)] | 90 days
  Proctitis as assessed using Common terminology criteria for adverse events (CTCAE)

SECONDARY OUTCOMES:
Cystitis [assessed using CTCAE Grading Criteria] | 90 days
  Cystitis as assessed using CTCAE Grading Criteria
Hematologic Toxicity | 90 days
  Hematologic Toxicity as assessed by significant reduction in hematologic components
Biochemical progression-free survival (b-PFS) | 5-years
  b-PFS as assessed using Prostate-Specific Antigen (PSA)
Treatment Response | 3 months after treatment termination
  Treatment Response as assessed using Magnetic Resonance Imaging techniques

CONTACTS AND LOCATIONS:
Overall Officials: Abolfazl Razzaghdoust, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shohada-e-Tajrish Medical Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No